CLINICAL TRIAL: NCT02941315
Title: EARLY Risk Stratification in CardioMYOpathies With Unknown Etiology for Heart Failure
Brief Title: Risk Stratification of Heart Failure in Cardiomyopathies.
Acronym: EARLY-MYO-HF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015015K
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2022-11

CONDITIONS: Cardiomyopathy With Unknown Etiology
Keywords: Cardiomyopathy; Heart Failure; Cardiac Magnetic Resonance
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Captopril; Adrenergic beta-Antagonists; Furosemide; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- with CMR confirmed etiology (Experimental): Participants who were identified with cardiac magnetic resonance (CMR) in etiology were treated with drug including etiologic treatment,anti-myocardial remodeling.
  Interventions: Drug: etiologic treatment,anti-myocardial remodeling
- etiology unconfirmed without acute HF (Placebo Comparator): Participants who were not identified with cardiac magnetic resonance (CMR) in etiology and without acute hearts failure (HF) were treated with drug with anti-myocardial remodeling.
  Interventions: Drug: anti-myocardial remodeling
- etiology unconfirmed with acute HF (Placebo Comparator): Participants who were not identified with CMR in etiology but with acute hearts failure were treated with drug with anti-myocardial remodeling,anti-acute heart failure.
  Interventions: Drug: anti-myocardial remodeling,anti-acute heart failure
- etiology confirmed with acute HF (Experimental): Participants who were identified with CMR in etiology but with acute hearts failure were treated with drug with Etiological, anti-remodeling and symptom treatment.
  Interventions: Drug: Etiological, anti-remodeling and symptom treatment

INTERVENTIONS:
Drug: etiologic treatment,anti-myocardial remodeling — When the etiology was diagnosed clearly by cardiac magnetic resonance(CMR), participants were treated with drugs including etiologic treatment,anti-myocardial remodeling according to guidelines for treatment of cardiomyopathy.
  Other Names: Etiology treatment, captopril, beta-blocker
  Arms: with CMR confirmed etiology
Drug: anti-myocardial remodeling — When the etiology was not diagnosed clearly by cardiac magnetic resonance(CMR), in participant without companioned with acute heart failure, participants were treated with drugs including anti-myocardial remodeling according to guidelines for treatment of cardiomyopathy.
  Other Names: Captopril, beta-blocker
  Arms: etiology unconfirmed without acute HF
Drug: anti-myocardial remodeling,anti-acute heart failure — When the etiology was not diagnosed clearly by cardiac magnetic resonance(CMR), in participant companioned with acute heart failure, participants were treated with drugs including anti-myocardial remodeling and anti- acute failure according to guidelines.
  Other Names: captopril, fursemide, spironolactone
  Arms: etiology unconfirmed with acute HF
Drug: Etiological, anti-remodeling and symptom treatment — When the etiology was diagnosed clearly by cardiac magnetic resonance(CMR), in participants were companioned with acute heart failure, the participant should be treated with drugs including etiologic treatment,anti-myocardial remodeling and anti-acute heart failure according to guidelines for treatment of cardiomyopathy.
  Other Names: Etiology treatment,captopril, fursemide, spironolactone
  Arms: etiology confirmed with acute HF

SUMMARY:
The investigators aimed to use CMR technique in helping diagnose the etiology of unknown cardiomyopathy. Try to make a risk stratification of susceptible heart failure based on the extent of myocardial impairment.

DETAILED DESCRIPTION:
Cardiomyopathy is a category of multiple causes of myocardial injury in structure and function, of which unexplained cardiomyopathy was most worried by cardiologists. Since the etiology confirmation sometimes still lacks of effective tools, therefore it can not be treated against etiology and may gradually developing to systolic or diastolic heart failure. The development of heart failure can be in different speeds, varying degrees, inconsistent in reversibility, and distinct response to treatment of heart failure.

In "real-world", ECG , cardiac ultrasound and myocardial enzymology can not be the whole to indicate the etiology of heart failure, so a strong clinical tool in the existing auxiliary examination is urgently needed and help to assess the risk of potential heart failure, therefore a reasonable treatment time window can be proposed.

The investigators aimed to use CMR technique in helping diagnose the etiology of unknown cardiomyopathy. Try to make a risk stratification of susceptible heart failure based on the extent of myocardial impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cardiomyopathy diagnosed by medical history, clinical symptoms, laboratory tests including ECG, echocardiography.
* no known etiology of cardiomyopathy was confirmed.

Exclusion Criteria:

* with contraindications of magnetic resonance include: 1, participants with cardiac pacemakers and nerve stimulator; 2, participants who have done aneurysm surgery and intracranial with aneurysm folder; 3, participants with the metal foreign body in the eye; 4, pregnant women; 5, critically ill participants need life support systems; 6, epilepsy participants; 7, claustrophobic participants;.
* participants who are <15 years of age or >75 years.
* participants who have the contraindication use of contrast media: glomerular filtration rate <30 ml/min

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
hospitalization due to heart failure | 6 months after the first visit
  Evaluate the relationship between scar amount and hospitalization due to heart failure

SECONDARY OUTCOMES:
malignant arrythmia | 6 months after the first visit
  Evaluate the relationship between scar amount and malignant arrythmia
mortality | 6 months after the first visit
  Evaluate the relationship between scar amount and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No